CLINICAL TRIAL: NCT00256048
Title: Efficacy of Nasojejunal Enteral Feeding in Critically Ill Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Melbourne Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002.228
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2015-04

CONDITIONS: Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Patients will receive enteral nutrition via a nasogastric tube as per standard feeding regime
- Nasojejunal Arm (Active Comparator): Patient will receive feeding via a nasojejunal feeding tube
  Interventions: Procedure: Nasojejunal feeding

INTERVENTIONS:
Procedure: Nasojejunal feeding
  Arms: Nasojejunal Arm

SUMMARY:
The purpose of this study is to determine if naso-jejunal feeding (feeding beyond the stomach) improves the efficacy of enteral feeding (feeding into the gut) in critically ill patients.

The study hypothesis is that in patients who fail to establish enteral feeding via the nasogastric route, introduction of nasojejunal feeding will lead to more effective enteral feeding than the current regime involving staged introduction of promotility agents.

DETAILED DESCRIPTION:
The study examines the area of enteral feeding in critically ill patients. Current standard enteral feeding practice is via a nasogastric with the addition of promotility agents for patients who fail to absorb their enteral nutrition.

This study compares the efficacy of nasojejunal feeding feeding with nasogastric enteral feeding with the addition of promotility agents.

The duration of feeding will be determined by the patients nutritional requirements and their general condition. However the data will be collected for duration of enteral feeding, 28 days or ICU discharge whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18years or over) admitted to the ICU with an expected stay of more than 48 hours.
2. Patients commenced on enteral feeding via a nasogastric tube who fail to tolerate gastric feeding due to excessive gastric aspirate volumes.
3. Patients who consent or if the patient is incompetent, the next of kin, who consent, to inclusion in the study.

   -

Exclusion Criteria:

1. patients less than 18 years of age.
2. Patients with known allergy to promotility agents, metoclopramide or erythromycin.
3. Patients with a contra indication to nasojejunal feeding. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-05; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of feeding | participants will be followed until death, discharge from ICU, commencement of oral or parental nutrition or 28 days post ICU admission

SECONDARY OUTCOMES:
1. To determine the incidence of complications with enteral feeding via nasogastric and nasojejunal routes. | participants will be followed until death, discharge from ICU, commencement of parental or oral nutrition or 28 days post ICU admission.
2. To assess the efficacy of current strategies for optimising enteral feeding efficacy. | participants will be followed until death, discharge from ICU commencement of oral or parental nutrition,or 28 days post ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Robertson, Principal Investigator — Intensive Care Unit, Royal Melbourne Hospital
Locations (1):
- Intensive Care Unit, Royal Melbourne Hospital, Grattan Street, Parkville, Victoria, Australia